CLINICAL TRIAL: NCT03054311
Title: Lifestyle Matters: An Occupational Approach Towards Health and Well-being in Later Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Responsible Party: Principal Investigator, Professor Gail Mountain, Professor of Health Services Research (assisted living research), University of Sheffield
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2006/01/GM
Record Dates: First submitted 2017-01-19; First posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Mental Health Wellness 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle Matters intervention (Experimental)
  Interventions: Behavioral: Lifestyle Matters

INTERVENTIONS:
Behavioral: Lifestyle Matters

SUMMARY:
Lifestyle Matters is an occupational approach to healthy ageing, which helps older people to get the most out of life. The intervention is based on an American model of health promotion called Lifestyle Redesign. This was found to be highly effective in enhancing the physical and mental health, occupational functioning and life satisfaction of community living older adults in Los Angeles, USA.

Weekly group meetings provide older people with the space, time and opportunity to share their experiences. Through a process of peer exchange and guidance, participants have the opportunity to reflect upon the range of activities that they engage with. They are then helped to begin to understand how these activities might impact on their health and well-being. However this approach alone cannot meet the complex needs of individual older people, and their specific and personal concerns. In recognition of this, the programme also includes monthly individual sessions with one of the group facilitators. The older person in partnership with the facilitator identifies a tailored programme to meet their individual needs, including the means by which they might work towards their personal goals. The individual programme is updated and refreshed in subsequent meetings over the months.

During 2004/5 researchers at Sheffield Hallam University in partnership with other researchers in York and Leeds, and clinical colleagues in Sheffield explored the feasibility of delivering this intervention to older people living in the UK. The project was funded through the Sheffield Health and Social Research Consortium. The summary below is an account of the process and outcomes of delivering a Lifestyle Matters programme to two groups of community living older people during 2004/5.

ELIGIBILITY:
Inclusion Criteria:

* Community living
* Aged 65 or over

Exclusion Criteria:

* Score of 18 or under on Mini-Mental State Examination (MMSE)
* high level of depression, assessed using the Geriatric depression rating scale (GDS)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-01; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Mini Mental State examination | On average 8 months after commencing intervention

SECONDARY OUTCOMES:
Geriatric Depression Rating Scale | On average 8 months after commencing intervention
Barthel Index | On average 8 months after commencing intervention
SF36 Quality of Life | On average 8 months after commencing intervention
WHODAS (World Health Disability Assessment Schedule) | On average 8 months after commencing intervention
Nottingham Leisure Questionnaire | On average 8 months after commencing intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Hallam University, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mountain GA, Craig CL. The lived experience of redesigning lifestyle post-retirement in the UK. Occup Ther Int. 2011 Mar;18(1):48-58. doi: 10.1002/oti.309. Epub 2010 Dec 9. PMID 21341343
- [Derived] Chatters R, Newbould L, Sprange K, Hind D, Mountain G, Shortland K, Powell L, Gossage-Worrall R, Chater T, Keetharuth A, Lee E, Woods B. Recruitment of older adults to three preventative lifestyle improvement studies. Trials. 2018 Feb 20;19(1):121. doi: 10.1186/s13063-018-2482-1. PMID 29458392